CLINICAL TRIAL: NCT06943014
Title: Development and Validation of an Actimetric Protocol to Quantify Physical Activity and Sedentary Behaviour in Post-stroke Subjects
Acronym: ActiStroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025/11FEV/062
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Chronic Stroke Patients; Stroke With Hemiparesis
Keywords: Physical activity monitoring; Stroke rehabilitation; Actimetry; Accelerometers; Pressure insoles; Energy expenditure estimation; Inactivity tracking; Actimetry to measure physical activity and sedentary behavior in stroke patients
MeSH Terms: conditions — Stroke | interventions — Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actimetry protocol (Experimental): All participants follow the same actimetry-based monitoring protocol. There are no comparison groups or randomized interventions. Therefore, the study includes only one arm. Participants will wear motion sensors (accelerometers and pressure insoles) to quantify physical activity and sedentary behavior.
  Interventions: Device: Actimetry Protocol

INTERVENTIONS:
Device: Actimetry Protocol — Our goal is to develop an actimetry protocol using both accelerometers and pressure insoles to quantify physical activity, involving the upper and/or lower limbs, as well as sedentary behavior in post-stroke individuals. Recent studies have explored the use of validated accelerometer configurations designed for healthy individuals, applied to the post-stroke population to monitor their physical activity and sedentary behavior. However, although these protocols have been validated for healthy individuals, they need to be adapted for post-stroke patients, who exhibit slower, asymmetric, and lower-amplitude movements compared to healthy subjects. This protocol could be valuable in both clinical practice and research, helping to optimize stroke rehabilitation and promote a healthy, active lifestyle.
  Other Names: Accelerometry; Accelerometer

SUMMARY:
The aim of this project is to develop an actimetry protocol based on a system of motion sensors, such as accelerometers and pressure insoles.

These sensors will be used to analyze arm and leg movements in individuals who have experienced a stroke. Throughout the study, the investigators will adjust certain parameters-such as sensor placement and measurement frequency-to optimize data quality.

They will also refine data analysis methods to better identify the types of movements performed (upper and lower limbs), estimate energy expenditure, and recognize different postures adopted by the participant (sitting, standing, etc.).

The goal of this protocol is to provide accurate measurements of physical activity and inactivity, both in controlled environments (such as a laboratory) and in real-life settings (outdoors or at home).

This study will allow us to validate the reliability of the actimetry protocol and assess how easy it is to use at home.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Stroke diagnosed by a neurologist and confirmed by medical imaging
* More than 14 days post-stroke
* Medically stable condition
* Hemiparesis with impaired locomotion: Functional Ambulation Classification (FAC) between 1 and 5
* Montreal Cognitive Assessment (MoCA) score > 18/30

Exclusion Criteria:

* Inability to understand simple instructions
* Other neurological or musculoskeletal disorders limiting functional mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Actimetry protocol | By the completion of the home monitoring phase, expected around April 2027
  Development of an actimetry protocol using accelerometers and pressure insoles for post-stroke subjects.

SECONDARY OUTCOMES:
Validation, feasibility, and usability of the actimetry protocol across different environments | By the completion of the home monitoring phase, expected around April 2027
  Validation of an actimetry protocol in the post-stroke population in a controlled environment (laboratory), in an ecological setting (outdoor), and assessment of its feasibility and usability at home.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium